CLINICAL TRIAL: NCT01017003
Title: An Open Label, Two Period, Sequential, Single Dose and Multiple Dose Pharmacokinetic Study With 0.6mg Colchicine Tablets in Healthy Volunteers
Brief Title: Pharmacokinetic Study With Colchicine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-07-1004
Record Dates: First submitted 2009-08-13; First posted 2009-11-20 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: healthy; pharmacokinetics
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 0.6mg colchicine tablet
  Interventions: Drug: colchicine tablets
- 2 (Experimental): colchicine 0.6mg q12 hours for 10 days
  Interventions: Drug: colchicine tablets

INTERVENTIONS:
Drug: colchicine tablets — 0.6mg colchicine tablet
  Other Names: COLCRYS TM
  Arms: 1
Drug: colchicine tablets — 0.6mg q12 hours for 10 days
  Other Names: COLCRYS TM
  Arms: 2

SUMMARY:
This open label, single group, sequential dose study will compare the single dose pharmacokinetics of colchicine 0.6 mg given orally to colchicine pharmacokinetics after 10 days of a standard prophylactic dose (0.6 mg every 12 hours) in healthy volunteers.

DETAILED DESCRIPTION:
This open label, single group, sequential dose study will compare the single dose pharmacokinetics of colchicine 0.6 mg given orally to colchicine pharmacokinetics after 10 days of a standard prophylactic dose (0.6 mg every 12 hours) in healthy volunteers. After a fast of at least 10 hours, fourteen healthy non-smoking, non-obese, non-pregnant volunteers will receive a single oral dose of colchicine 0.6 mg. Fasting will continue for 4 hours after the dose, at which time a standard meal will be served. Blood will be drawn from all participants at times sufficient to adequately define the single dose pharmacokinetics of colchicine and its 3 major metabolites, 2, 3 and 10 demethylcolchicine. Following a 14 day washout period, all participants will begin a 10 day regimen of colchicine 0.6 mg orally every 12 hours. On the morning of day 25, after a fast of at least 10 hours, all participants will receive their final dose of colchicine 0.6 mg. Again blood will be drawn at times sufficient to determine the pharmacokinetics of colchicine and its 3 major metabolites after chronic dosing. The pharmacokinetic parameters for each dosing situation will be derived and compared for relevant differences. Though not a specific goal of this study, all participants will be monitored for adverse events by observation and query during periods of confinement on days 1, 15 and 25, as well as by complete blood count (CBC) with differential and clinical chemistry, sitting and standing blood pressures, and heart rate and 12-lead electrocardiogram (EKG) before and after dosing, on days 1 and 25.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the screening process within 28 days prior to Period I dosing
* Healthy non-smoking, non-obese adult men and women volunteers between the ages of 18 to 45 years of age, weighing at least 110 with a body mass index of 18-30kg/m2
* Women must be postmenopausal, surgically sterile, commit to abstinence from heterosexual sexual contact or use two methods of contraception.

Exclusion Criteria:

* Pregnant or lactating
* Use of any investigational drug within 28 days prior to Period I dosing.
* Presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the clinical investigator(s)
* Positive screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Clinical laboratory test values outside the accepted reference range and when confirmed on re-examination.
* Any clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators)
* Use of any systemic prescription medication in the 14 days prior to Period I dosing
* History of any allergy(s) including allergy to colchicine or related drugs.
* History of drug or alcohol addiction or abuse within the past year or a positive drug abuse screen
* Currently or recent (within 6 months) use of tobacco products prior to dose administration
* Donation of greater than 150 mL of blood within 28 days or plasma within 14 days prior to period I dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS Institiute, Ltd.
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Colchicine - Single Dose, Twice Daily Dose, Final Single Dose: All subjects received a single dose of colchicine 0.6 mg on Day 1 following an overnight fast. After a 14-day washout period, subjects received colchicine 0.6 mg every 12 hours for 10 days. On the morning of Day 25, subjects received their final colchicine 0.6 mg dose following an overnight fast.
Period: Single Dose Colchicine 0.6 mg, Day 1
Arm/Group | Colchicine - Single Dose, Twice Daily Dose, Final Single Dose
Started | 13
Completed | 13
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine - Single Dose, Twice Daily Dose, Final Single Dose
Started | 13
Completed | 13
Not Completed | 0
Period: Colchicine 0.6 mg Twice Daily x 10 Days
Arm/Group | Colchicine - Single Dose, Twice Daily Dose, Final Single Dose
Started | 13
Completed | 13
Not Completed | 0
Period: Colchicine 0.6 mg Final Dose
Arm/Group | Colchicine - Single Dose, Twice Daily Dose, Final Single Dose
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine - Single Dose, Twice Daily Dose, Final Single Dose
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 25.5 [19 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: maximum serum concentration measured after a single oral dose in fasted healthy adults and after a single oral dose in fasted healthy adults at steady state for comparison of the two conditions
Time Frame: Pharmacokinetic samples collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing
Population: per protocol
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Pharmacokinetics (Day 1): 0.6mg colchicine orally administered to healthy fasted volunteers as a single isolated dose (Day 1)
- Colchicine Pharmacokinetics at Steady State (Day 25): 0.6mg colchicine tablet administered to healthy fasted volunteers after a regimen of oral colchicine 0.6mg every 12 hours for 10 days (Day 25)
Arm/Group | Colchicine Pharmacokinetics (Day 1) | Colchicine Pharmacokinetics at Steady State (Day 25)
Number analyzed (Participants) | 13 | 13
pg/mL | 2450.15 (702.11) | 3553.15 (843.45)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to the Time of the Last Measured Level.
Description: Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (t), calculated using the linear trapezoidal rule.
Time Frame: 0.0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 36, 48, 72, and 96 hours after dosing
Population: by protocol
Measure: Mean (Standard Deviation); unit: pg-h/ml
Arm/Group | Colchicine Pharmacokinetics (Day 1) | Colchicine Pharmacokinetics at Steady State (Day 25)
Number analyzed (Participants) | 13 | 13
pg-h/ml | 10494.66 (3544.08) | 43576.96 (9333.26)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC 0-inf)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: 0.0, 0.5, 1,1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing
Population: by protocol
Measure: Mean (Standard Deviation); unit: pg-h/ml
Arm/Group | Colchicine Pharmacokinetics (Day 1) | Colchicine Pharmacokinetics at Steady State (Day 25)
Number analyzed (Participants) | 13 | 13
pg-h/ml | 12268.18 (4422.08) | 54198.77 (9214.54)

ADVERSE EVENTS:
Arm/Group | Colchicine Pharmacokinetics (Day 1) | Colchicine Pharmacokinetics at Steady State (Day 25)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Pharmacokinetics (Day 1) | Colchicine Pharmacokinetics at Steady State (Day 25)
Diarrhea (Gastrointestinal disorders) | 0/13 (0) | 1/13 (1)
Dry Mouth (Gastrointestinal disorders) | 0/13 (0) | 1/13 (1)
Stomach Discomfort (Gastrointestinal disorders) | 0/13 (0) | 1/13 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0/13 (0) | 1/13 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0/13 (0) | 1/13 (1)
Dizziness (Nervous system disorders) | 0/13 (0) | 1/13 (1)

LIMITATIONS AND CAVEATS:
14 subjects were sought, 13 enrolled due difficult recruitment. It was impossible to determine the kinetics of metabolites because none reached the level of detectability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days